CLINICAL TRIAL: NCT04471129
Title: Non-invasive Ventilation and High-speed Oxygen Therapy Effects on Heart Function - HiFlow-Heart Study
Acronym: HiFlow-Heart
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019/0400/HP
Record Dates: First submitted 2020-06-25; First posted 2020-07-15 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-06

CONDITIONS: Chronic Heart Failure
Keywords: chronic heart failure; heart surgery; invasive mechanical ventilation; high flow oxygen therapy

STUDY DESIGN:
Intervention Model Description: sequential assignment
Masking Description: No applicable
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Flow Oxygen Therapy, followed by Non-Invasive Ventilation (Other): oxygenation first by High-Flow Oxygen Therapy, then by O2C, then by Non-Invasive Ventilation
  Interventions: Other: HFO/O2C/NIV
- Non-Invasive Ventilation, followed by High-Flow Oxygen Therapy (Other): oxygenation first by Non-Invasive Ventilation, then by O2C, then by High-Flow Oxygen Therapy
  Interventions: Other: NIV/O2C/HFO

INTERVENTIONS:
Other: HFO/O2C/NIV — High-flow oxygen therapy + O2C + Non invasive ventilation
  Arms: High-Flow Oxygen Therapy, followed by Non-Invasive Ventilation
Other: NIV/O2C/HFO — Non invasive ventilation + O2C + High-flow oxygen therapy
  Arms: Non-Invasive Ventilation, followed by High-Flow Oxygen Therapy

SUMMARY:
The investigators hypothesize that the airway pressures generated by High Flow Oxygen Therapy could have a beneficial impact in patients with heart failure, particularly by lowering capillary pulmonary arterial pressures. However, results compared to Non-Invasive Ventilation are difficult to predict due to the lack of data in the literature.

DETAILED DESCRIPTION:
The investigators propose to carry out a prospective randomized cross-over prospective physiological study comparing, Non-Invasive Ventilation and High Flow Oxygen Therapy in patients with chronic uncompensated heart failure. This stable population would make it possible to easily study variations in a physiological parameter without any added risk for the patient, but with all the pathophysiological parameters transposable to the situation of decompensated heart failure.

Indeed, it is accepted that the existence of heart failure with decreased left ventricular ejection fraction (LVEF) (< 40%) exposes patients to a high risk of congestive cardiac decompensation due to the associated presence of diastolic dysfunction1.

The study will be conducted using an alternating design, where a patient receives the two treatments one after the other ("cross-over"), because the alternating design, compared to the two parallel arm design, reduces the number of patients needed to show a given difference between High Flow Oxygen Therapy and Non-Invasive Ventilation at equal power, if there is neither an order-of-prescription effect ("period") nor a residual effect of the first treatment on the second treatment ("carry-over"). In order to avoid a residual effect on changes in pressure or oxygenation, a wash-out period on conventional oxygen therapy (O2C) should be set between the two treatments (High Flow Oxygen Therapy and Non-Invasive Ventilation) administered to the same patient.

ELIGIBILITY:
Inclusion Criteria:

1. Major patient
2. Patient who has undergone cardiac surgery with extracorporeal circulation for more than 24 hours and has been extubated for at least 6 hours.
3. Pre-operative heart failure with left ventricular ejection fraction < 40%.
4. Invasive monitoring by pulmonary arterial catheter (Swan-Ganz) with transpulmonary thermodilution and by radial arterial catheter intended for use in the intra- and post-operative monitoring of the patient.
5. Treatment with conventional oxygen therapy (O2C) without an increase in O2 flow for more than 30 minuts, without signs of hypoxemia (SpO292%)
6. Stable hemodynamic parameters: no changes in hemodynamic parameters (arterial pressures and pulmonary and cardiac index) by more than 10% over the 30 minutes prior to inclusion and no increase in cardiotropic medication for at least 30 minutes.
7. Patient with an oxygenation rate ≤ 6L
8. For women of child-bearing age: negative pregnancy test at inclusion
9. Person who has read and understood the information letter and signed the consent form
10. Affiliation to a social security scheme

Exclusion Criteria:

1. Contraindication to the use of NIV or HFO
2. Patient with orotracheal intubation or tracheotomy
3. Renal failure with hemodialysis or hemofiltration
4. Uncontrolled state of shock (PAS<90 mmHg and/or cardiac index<1.8 L/min/m² and/or norepinephrine>0.2 μg/kg/min and/or dobutamine>10 μg/kg/min)
5. Acute respiratory failure as defined by :

   * clinical signs: respiratory rate >35/min, signs of struggle, SpO2<92% on O2C
   * indication for treatment with NIV or HFO at the discretion of the clinician
   * oxygen dependency requiring O2C>6L/min O2C flow at the oxygen mask
6. Chronic advanced respiratory disease
7. Chronic treatment with NIV or CPAP at home
8. Non-operated aortic or mitral insufficiency ≥ II/IV
9. Administration of loop diuretics within 3 hours prior to inclusion for intravenous forms and within 6 hours for oral forms.
10. Presence of altered consciousness defined by a Glasgow score < 15/15 or cognitive dysfunction defined by a CAM-ICU score > 0/4
11. Pregnant or parturient or nursing woman or proven lack of effective contraception
12. Person deprived of liberty by an administrative or judicial decision or person placed under judicial protection / subtutorship or guardianship
13. Person participating in another trial / having participated in another trial that may interfere with the procedures that are the subject of the research within a 4-week time frame

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-07-15 (Estimated); Primary Completion 2022-07-15 (Estimated); Study Completion 2022-10-15 (Estimated)

PRIMARY OUTCOMES:
High-Flow Oxygen Therapy and Non Invasive Ventilation on left ventricular filling pressures | Day 1
  Difference between High-Flow Oxygen Therapy and Non Invasive Ventilation on left ventricular filling pressures as assessed by the occluded pulmonary artery occlusion pressure (in mmHg) measured by Swan-Ganz pulmonary artery catheterization

SECONDARY OUTCOMES:
Comparison between High-Flow Oxygen Therapy and Non-Invasive ventilation w.r.t. ventricular function | Day 1
  Arterial pressure [mmHg] measured by Swan-Ganz catheter
Comparison between High-Flow Oxygen Therapy and Non-Invasive ventilation w.r.t. arterial oxygenation | Day 1
  Arterial oxygen saturation, SaO2 [%], measured by Swan-Ganz catheter
Comparison between High-Flow Oxygen Therapy and Non-Invasive ventilation w.r.t. change in pulmonary volume | Day 1
  End-expiratory lung impedance (mean of 3 measures), measured by PulmoVista (Draeger, Germany)
Patient comfort | Day 1
  Patient's evaluation of comfort on Visual Analog Scale (10 points)